CLINICAL TRIAL: NCT06840340
Title: Effects of Concurrent Activiation Potentation Induced by Customized Mouth Guard on Baseball and Softball Performance
Brief Title: Customised Mouthguards on Baseball and Softball Performance
Acronym: CM&Baseball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114-1; 114-1 (Other: NTUS)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Oral Manifestations; Control Condition
Keywords: concurrent activation potentiation; bite force
MeSH Terms: conditions — Oral Manifestations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mouthguards (Experimental): Participants wore the mouthguard
  Interventions: Device: Customised mouthguards
- Control (No Intervention): Participants did not ware the mouthguard

INTERVENTIONS:
Device: Customised mouthguards — Wore customised mouthguards and measurement athletic performance of baseball and softball performance.
  Arms: Mouthguards

SUMMARY:
Whether the use of customised mouthguards is effective in improving the athletic performance of baseball and softball performance

DETAILED DESCRIPTION:
This study recruited 45 baseball and softball players, including 30 fielders and 15 pitchers. Using a randomized crossover experimental design, the study was divided into randomised divided into customised mouthguards trial (MG) and control trial (CON) without temporal positioning. After the participants wore the mouthguard, they performed the vertical jump and grip strength tests sequentially. At the end of the test, depending on the pitcher or fielder, a baseball pitching ability test or a hitting ability test was conducted using a radar baseball tracking system. It is expected to analyze the vertical jump height, grip strength, pitchers' straight and changeup ball speeds, rotation speeds, degree of displacement, on-base and off-base locations. Hitting ability was expected to be documented with respect to initial velocity, elevation, and consistency of elevation.

ELIGIBILITY:
Inclusion Criteria:

* has won the top 8 national level baseball of softball championships in the last three years.
* no cardiovascular and joint diseases.
* aged 20 or above who are adults
* continuing to train professionally more than 5 days a week for the past year

Exclusion Criteria:

* have not won the top 8 national baseball or softball championships in the past three years.
* have a cardiovascular or joint disease, or any injuries that may be impaired by exercise.
* participants who are underage or not in regular baseball or softball training
* have injury to the temporomandibular joint.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
exit velocity | Immediately after wore customized mouthguard or not
  Test the pitching or batting exit velocity

CONTACTS AND LOCATIONS:
Overall Officials: Chih Hui Chiu, PhD, Principal Investigator — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, North, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan

REFERENCES:
- [Derived] Teng NC, Hu YH, Wu TI, Shiu YJ, Yen CW, Chan WJ, Chiu CH. Biting on Customized Mouthguards Improves Vertical Jump and Slider Quality of Baseball Pitchers. J Strength Cond Res. 2025 Aug 13. doi: 10.1519/JSC.0000000000005233. Online ahead of print. PMID 40845272

DOCUMENTS (1):
  • Study Protocol (2025-02-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT06840340/Prot_000.pdf